CLINICAL TRIAL: NCT02563691
Title: Comprehensive Stereotactic Radiotherapy for Oligometastatic Prostate Cancer: A Phase I/II Study
Brief Title: Stereotactic Radiotherapy for Oligometastatic Prostate Cancer
Acronym: CROP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Patrick Cheung, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROP
Record Dates: First submitted 2015-07-03; First posted 2015-09-30 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Stereotactic radiotherapy will be delivered to the prostate (if not previously treated) and to all metastatic tumours.
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy — Patients will receive ADT for a minimum of 1 year. After this, an intermittent hormone therapy approach will be taken.
  The prostate (if not previously treated) will be treated to a dose of 35-40 Gy in 5 fractions. All visible nodal metastases will be treated to a dose of 30-35 Gy in 5 fractions. Non-spine bone metastases will be treated to a dose of 30-40 Gy in 5 fractions. Metastases in the brain, spine, lung, liver, and adrenal will be treated according to established SRT policies at the Sunnybrook Odette Cancer Centre. Comprehensive SRT should be delivered within 3 months of starting ADT.
  Other Names: SBRT, SABR

SUMMARY:
This is a study that assesses the safety and efficacy of using stereotactic radiotherapy in conjunction with hormone therapy for patients with metastatic prostate cancer where there are a limited number of metastatic tumours.

DETAILED DESCRIPTION:
Patients will receive androgen deprivation therapy (ADT) for a minimum of 1 year. After this, an intermittent hormone therapy approach will be taken, where ADT will not be restarted until the prostate specific antigen (PSA) reaches a minimum of 10-15 ng/mL. Lupron 30 mg IM will be delivered every 4 months when on ADT.

The prostate (if not previously treated) will be treated to a dose of 35-40 Gy in 5 fractions. All visible nodal metastases will be treated to a dose of 30-35 Gy in 5 fractions. It is very likely that nodal metastases will shrink significantly (often completely) with ADT. In this scenario, the involved nodal regions will be treated to a more modest dose of 25 Gy in 5 fractions (roughly equivalent to a dose of 46 Gy in 23 fractions assuming an α/β value of 1.4). Non-spine bone metastases will be treated to a dose of 30-40 Gy in 5 fractions. Metastases in the brain, spine, lung, liver, and adrenal will be treated according to established stereotactic radiotherapy (SRT) policies at Sunnybrook Odette Cancer Centre. Comprehensive SRT should be delivered within 3 months of starting ADT.

During any "off" period of ADT (before the PSA rises above 10-15 ng/mL), comprehensive SRT can be repeated if there are new oligometastases that become visible. One month after initiation comprehensive SRT, patients will be contacted to assess for acute toxicities.

After completion of radiotherapy to all disease sites, patients will be followed every 3-4 months with PSA testing until the development of castrate resistant prostate cancer. At the same time points, late toxicity and quality of life will be collected for a minimum of 2 years. Computed tomography (CT) of the chest/abdo/pelvis +/- magnetic resonance imaging (MRI) of previously irradiated body sites and bone scan will be performed whenever the PSA reaches ≥ 10 ng/mL (prior to re-starting androgen deprivation therapy during intermittent hormone therapy approach), or at a minimum frequency of once per year.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* ECOG performance status 0-1.
* Histologic confirmation of prostate adenocarcinoma.
* Stage IV disease, with up to 5 metastatic tumours outside of the prostate and pelvic lymph nodes.
* ≤ 3 tumours within any given organ system (e.g. up to 3 brain metastases, or 3 liver metastases).
* All sites of disease are amenable to stereotactic radiotherapy.

Exclusion Criteria:

* Castrate resistant prostate cancer.
* Evidence of spinal cord compression.
* Previous radiotherapy for current cancer (with the exception of upfront management of the primary prostate tumour, brain metastasis(es) prior to androgen deprivation therapy).
* Inability to safely treat all sites of visible disease.
* Prior malignancy within the past 5 years, excluding non-melanoma skin cancer, and in-situ cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of late radiotherapy toxicities after stereotactic radiotherapy to all sites of disease | cumulative incidence at 2 years
  common terminology criteria for adverse events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Quality of Life (EORTC QLQ-C30) | proportion of patients who experience a significant decline in quality of life at 6 months, 12 months, 18 months, and 24 months
Time to development of castrate resistant prostate cancer | through study completion, an average of 2 years
Radiographic local control of irradiated tumours | actuarial rate at 2 years
Radiographic "distant" control rate | actuarial rate at 2 years
Overall survival | through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cheung, M.D., Principal Investigator — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada